CLINICAL TRIAL: NCT01467583
Title: Use of Fondaparinux in Critically Ill Patients With Renal Failure
Brief Title: Fondaparinux in Critically Ill Patients With Renal Failure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wayne State University (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Steven Dov Tennenberg, MD, Director, Surgical Intensive Care Unit, Wayne State University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 112050
Record Dates: First submitted 2011-11-03; First posted 2011-11-08 (Estimated); Results first posted 2015-06-19 (Estimated); Last update posted 2015-06-19 (Estimated); Status verified 2015-06

CONDITIONS: Venous Thromboembolism
Keywords: Fondaparinux; Renal Failure; Critically Ill
MeSH Terms: conditions — Venous Thromboembolism; Renal Insufficiency; Critical Illness | interventions — Fondaparinux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Renal failure on intermittent dialysis (Experimental): These are patients with renal failure, on intermittent hemodialysis (IHD), receiving fondaparinux 2.5 mg subcutaneously every 48 hours
  Interventions: Drug: Fondaparinux
- Renal failure-renal replacement therapy (Experimental): These are patients with renal failure, either acute or chronic, on continuous renal replacement therapy (CRRT) receiving fondaparinux 2.5 mg subcutaneously every 48 hours
  Interventions: Drug: Fondaparinux
- Renal failure, not on dialysis (Experimental): These are patients with acute kidney injury not yet on dialysis, receiving fondaparinux 2.5 mg subcutaneously every 48 hours
  Interventions: Drug: Fondaparinux

INTERVENTIONS:
Drug: Fondaparinux — 2.5 mg every 48 hours
  Other Names: Arixtra

SUMMARY:
The primary objective of this study is to determine whether a dose-adjusted prophylaxis fondaparinux regimen of 2.5 milligrams (mg) subcutaneously administered every (q) 48 hours (hr) in patients with renal failure achieves peak and trough levels similar to patients with normal renal function, and protects patients from developing venous thromboembolism (VTE). Our hypothesis is that a dose-adjusted fondaparinux regimen, which extends the dosing interval from q24 to q48 hr, in patients with estimated creatinine clearance of < 30 ml/min, will be safe and effective.

DETAILED DESCRIPTION:
We will be studying fondaparinux 2.5 mg subcutaneously every 48 hr in three distinct patient groups: 1) Acute kidney failure without hemodialysis, 2) Acute kidney failure (AKI) with intermittent hemodialysis (IHD) and 3) Acute renal failure with continuous renal replacement therapy (CRRT). All patients will be assessed for efficacy of the dose. Efficacy will be assessed by following clinically for any evidence of VTE, either deep venous thrombosis (DVT) or pulmonary embolism. In addition, lower extremity duplex studies will be performed at baseline and at the end of the study period to assess for DVT.

Secondary objectives will be safety and accumulation. Safety will be determined by assessment of clinically significant bleeding, defined as a drop in Hgb of > 2 grams (gm) in 24 hr, or the need for red blood cell transfusion related to bleeding. Accumulation may occur in renal failure and will be studied throughout the intensive care unit (ICU) stay through reevaluation of levels over time.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old and ≤ 89 years old
2. Body weight ≥ 50 kg or ≤ 150 kg
3. Estimated creatinine clearance of < 30 mL/min
4. Predicted ICU stay of more than 72 hours.

Exclusion Criteria:

1. Pregnant women
2. Infective Endocarditis
3. Neuraxial anesthesia or spinal puncture
4. Active bleeding
5. Treatment with vitamin K antagonists or therapeutic doses of unfractionated heparin
6. Signs of disseminated intravascular coagulation
7. Severe liver failure (serum bilirubin > 5 mg/dL)
8. Surgery planned within 24 hours of ICU admission
9. Latex allergy

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2011-11; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven D Tennenberg, MD, Principal Investigator — WSU, DMC
Locations (1):
- Detroit Medical Center, Detroit, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Renal Failure, on Intermittent Hemodialysis (IHD): These are patients with renal failure, on intermittent dialysis
  Fondaparinux: 2.5 mg every 48 hours
- Renal Failure, on CRRT on Fondaparinux: 2.5 mg Every 48 Hours: These are renal failure patients, either acute or chronic on Fondaparinux: 2.5 mg every 48 hours
- Renal Failure, Not on Dialysis Fondaparinux: 2.5 mg q48 hr: These are patients with acute kidney injury not yet on dialysis
  Fondaparinux: 2.5 mg every 48 hours
Period: Overall Study
Arm/Group | Renal Failure, on Intermittent Hemodialysis (IHD) | Renal Failure, on CRRT on Fondaparinux: 2.5 mg Every 48 Hours | Renal Failure, Not on Dialysis Fondaparinux: 2.5 mg q48 hr
Started | 16 | 4 | 12
Completed | 14 (Both patients completed > 1 dose and so their data was included in the results.) | 3 (Death unrelated to study drug on day #3. Data to that point is included in the results) | 10
Not Completed | 2 | 1 | 2
Not completed — Death | 1 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Renal Failure, on CRRT: Fondaparinux: 2.5 mg every 48 hours
- Renal Failure, Not on Dialysis: These are patients with acute kidney injury not yet on dialysis
  Fondaparinux: 2.5 mg every 48 hours
- Total: Total of all reporting groups
Arm/Group | Renal Failure, on Intermittent Hemodialysis (IHD) | Renal Failure, on CRRT | Renal Failure, Not on Dialysis | Total
Number analyzed (Participants) | 16 | 4 | 12 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (12) | 63 (10) | 62 (12) | 62 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 6 | 12
  Male | 11 | 3 | 6 | 20
Region of Enrollment [Number; unit: participants]
  United States | 16 | 4 | 12 | 32

OUTCOME MEASURES:

1. Primary Outcome: To Determine if an Adjusted-dose of Fondaparinux 2.5 mg Subcutaneously (SQ) q48 hr in Critically Ill Patients With Renal Failure Will Achieve Peak and Trough Levels Similar to Patients With Normal Renal Function on 2.5 mg SQ Daily Dosing of Fondaparinux.
Description: Fondaparinux Peak Levels measured at time +3 hours after the dose, and Trough Levels, measured at time + 47 hours post-dose around the first 5 doses of fondaparinux and then every 3rd dose thereafter. Levels will be sent to our hospital laboratory and performed using a calibrated fondaparinux assay.
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: mcg/ml
Groups:
- Renal Failure-continuous Renal Replacement Therapy: These are renal failure patients, either acute or chronic, on continuous renal replacement therapy (CRRT), receiving Fondaparinux: 2.5 mg every 48 hours
Arm/Group | Renal Failure, on Intermittent Hemodialysis (IHD) | Renal Failure-continuous Renal Replacement Therapy | Renal Failure, Not on Dialysis
Number analyzed (Participants) | 16 | 4 | 12
mcg/ml
  Peak Levels | 0.42 (0.16) | 0.31 (0.13) | 0.37 (0.21)
  Trough Levels | 0.18 (0.1) | 0.12 (0.09) | 0.17 (0.15)

2. Secondary Outcome: To Determine Number of Participants Who Experienced a Bleeding Event, Either Major or Minor, and to Determine the Number of Participants Who Experienced a Venous Thromboembolism During the Study Period
Description: Safety will be assessed through monitoring for clinical signs of bleeding. Major and minor bleeding will be documented. In additions, venous doppler studies of the bilateral lower extremities will be performed at study entry and study completion to monitor for any evidence of venous thromboembolism during the study period. We will report on the number of participants experiencing an adverse event during the study
Time Frame: 2 years
Measure: Number; unit: participants
Groups:
- Renal Failure on Intermittent Dialysis (IHD): These are patients with renal failure, on IHD, receiving fondaparinux 2.5 mg subcutaneously every 48 hours
  Fondaparinux: 2.5 mg every 48 hours
- Renal Failure-renal Replacement Therapy: These are patients with renal failure, either acute or chronic, receiving fondaparinux 2.5 mg subcutaneously every 48 hours
  Fondaparinux: 2.5 mg every 48 hours
Arm/Group | Renal Failure on Intermittent Dialysis (IHD) | Renal Failure-renal Replacement Therapy | Renal Failure, Not on Dialysis
Number analyzed (Participants) | 16 | 4 | 12
participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From study enrollment through until study discontinuation
Groups:
- Renal Failure-continuous Renal Replacement Therapy: These are patients with renal failure, on continuous renal replacement therapy (CRRT), receiving Fondaparinux: 2.5 mg every 48 hours
Arm/Group | Renal Failure, on Intermittent Hemodialysis (IHD) | Renal Failure-continuous Renal Replacement Therapy | Renal Failure, Not on Dialysis
Serious Adverse Events (participants affected / at risk) | 1/16 | 0/4 | 0/12
Other Adverse Events (participants affected / at risk) | 2/16 | 1/4 | 2/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Renal Failure, on Intermittent Hemodialysis (IHD) (N=16) | Renal Failure-continuous Renal Replacement Therapy (N=4) | Renal Failure, Not on Dialysis (N=12)
Clinically Significant Bleeding (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) — Number of patients who experienced clinically significant bleeding
Venous Thromboembolism (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) — Number of patients who experienced a venous thromboembolism
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Renal Failure, on Intermittent Hemodialysis (IHD) (N=16) | Renal Failure-continuous Renal Replacement Therapy (N=4) | Renal Failure, Not on Dialysis (N=12)
Minor Oozing (Minor Bleeding) (Blood and lymphatic system disorders) | 2 | 1 | 2 — Number of participants who experienced bleeding or oozing from lines, skin, hematuria, etc. None of these events were deemed clinically significant by the physician caring for the patient

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No